CLINICAL TRIAL: NCT01651052
Title: Clinical Trial of the Edwards Aortic Bioprosthesis, Model 11000
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-03
Record Dates: First submitted 2012-07-18; First posted 2012-07-26 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Aortic Valve Disorder; Aortic Valve Insufficiency; Aortic Valve Stenosis; Heart Failure; Coronary Artery Disease
Keywords: Aortic valve replacement/regurgitation
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Insufficiency; Aortic Valve Stenosis; Heart Failure; Coronary Artery Disease; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aortic Bioprosthesis, Model 11000 (Experimental): Aortic valve replacement therapy
  Interventions: Procedure: Heart Valve Surgery

INTERVENTIONS:
Procedure: Heart Valve Surgery — Implant of an aortic valve, Model 11000

SUMMARY:
The purpose of this observational trial is to gather further clinical data to confirm the safety and performance of the Edwards Pericardial Aortic Bioprosthesis, Model 11000 in this trial population.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, non-controlled observational clinical trial. Up to 200 subjects will be enrolled at up to 6 participating clinical sites. The trial will include male and female patients, 18 years or older, requiring replacement for a diseased, damaged, or malfunctioning native or prosthetic valve. Patients will be followed and assessed after implant for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Require replacement of aortic valve
* Signed informed consent
* Willing to return to study site for follow-up visits

Exclusion Criteria:

* Active endocarditis/myocarditis (< 3 months)
* Myocardial infarction (< 30 days)
* Renal insufficiency/ End-stage renal disease
* Life expectancy (< 1 year)
* Requires multiple valve replacement/repair
* Requiring emergent aortic valve surgery
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2011-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Sadowski, MD, Principal Investigator — John Paul II Hospital; Jacek Rozanski, MD, Principal Investigator — The Cardinal Stefan Wyszyński Institute of Cardiology
Locations (2):
- Poland (2):
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow
  - Instytut Kardiologii im. Prymasa Tysiąclecia Stefana Kardynała Wyszyńskiego, Warsaw

REFERENCES:
- [Background] De La Fuente AB, Wright GA, Olin JM, Duhay FG, Kapelak B, Bochenek M, Bartus K, Sadowski J. Advanced Integrity Preservation Technology Reduces Bioprosthesis Calcification While Preserving Performance and Safety. J Heart Valve Dis. 2015 Jan;24(1):101-9. PMID 26182627
- [Result] Bartus K, Litwinowicz R, Kusmierczyk M, Bilewska A, Bochenek M, Stapor M, Wozniak S, Rozanski J, Sadowski J, Kapelak B. Primary safety and effectiveness feasibility study after surgical aortic valve replacement with a new generation bioprosthesis: one-year outcomes. Kardiol Pol. 2018;76(3):618-624. doi: 10.5603/KP.a2017.0262. Epub 2018 Jan 3. PMID 29297188
- [Result] Sadowski J, Bartus K, Kapelak B, Chung A, Stapor M, Bochenek M. Aortic valve replacement with a novel anti-calcification technology platform. Kardiol Pol. 2015;73(5):317-22. doi: 10.5603/KP.a2014.0214. Epub 2014 Nov 5. PMID 25371311
- [Derived] Bartus K, Litwinowicz R, Bilewska A, Stapor M, Bochenek M, Rozanski J, Sadowski J, Filip G, Kusmierczyk M, Kapelak B. Final 5-year outcomes following aortic valve replacement with a RESILIA tissue bioprosthesis. Eur J Cardiothorac Surg. 2021 Jan 29;59(2):434-441. doi: 10.1093/ejcts/ezaa311. PMID 33141188

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 133 Subjects were enrolled and implanted with the study valve, for which data is available.
Period: Overall Study
Arm/Group | Aortic Bioprosthesis, Model 11000
Started | 133
Study Valve Group | 133
Completed | 107
Not Completed | 26
Not completed — Death | 21
Not completed — Explant | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 113
  Unknown or Not Reported | 20
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 133

OUTCOME MEASURES:

1. Primary Outcome: Number of Early Adverse Events Divided by Number of Subjects (Expressed as a Percentage)
Description: Number of early adverse events occurring within 30 days of procedure divided by the number of enrolled subjects times 100
Time Frame: Events occurring within 30 days of procedure
Measure: Number; unit: percentage
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
percentage
  All Cause Mortality | 2.3
  Trial valve-related Mortality | 0.8
  Study Valve Related Reoperation | 0.0
  Explant | 0.0
  Thromboembolism | 2.3
  Valve Thrombosis | 0.0
  Bleeding Event | 8.3
  Major Bleeding Event | 6.8
  Paravalvular Leak (PVL) | 0.8
  Major Paravalvular Leak | 0.0
  Endocarditis | 0.0
  Hemolysis | 0.0
  Nonstructural Valve Dysfunction (Not PVL) | 0.0
  Structural Valve Deterioration | 0.0

2. Primary Outcome: Number of Late Adverse Events Divided by Late Patient Years (Expressed as a Percentage)
Description: Number of late events divided by the total number of late patient years x 100. Late patient years are calculated from 31 days post-implant to the date of the last contact (follow up or adverse event).
Time Frame: Events occurring >= 31 days and up through 5 years post-implant
Measure: Number; unit: Percentage of events/late patient years
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
Percentage of events/late patient years
  All Cause Mortality | 3.2
  Trial valve-related mortality | 0.7
  Study Valve Related Reoperation | 0.2
  Explant | 0.2
  Thromboembolism | 0.4
  Valve Thrombosis | 0.2
  Bleeding Event | 0.4
  Major Bleeding Event | 0.4
  Paravalvular Leak (PVL) | 0.0
  Major Paravalvular Leak | 0.0
  Endocarditis | 0.2
  Hemolysis | 0.0
  Nonstructural Valve Dysfunction (Not PVL) | 0.2
  Structural Valve Deterioration | 0.0

3. Secondary Outcome: Subject's Average Mean Gradient Measurements
Description: Mean gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. Mean gradient values depend on the size and type of valve.
Time Frame: Baseline through 5-Year (at each scheduled follow-up visit)
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
mmHg
  Baseline | 49.4 (21.7)
  Discharge: number analyzed (Participants) | 130
  Discharge | 12.3 (5.3)
  3-6 months: number analyzed (Participants) | 128
  3-6 months | 12.2 (5.9)
  1 year: number analyzed (Participants) | 119
  1 year | 13.9 (6.1)
  2 year: number analyzed (Participants) | 110
  2 year | 13.8 (6.4)
  3 year: number analyzed (Participants) | 100
  3 year | 14.3 (6.1)
  4 year: number analyzed (Participants) | 98
  4 year | 15.0 (7.2)
  5 year: number analyzed (Participants) | 89
  5 year | 14.8 (7.6)

4. Secondary Outcome: Subject's Average Effective Orifice Area Measurements
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the aortic valve. Effective orifice area is evaluated by echocardiography over time.
Time Frame: Baseline through 5-Year (at each scheduled follow-up visit)
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: Centimeters squared
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
Centimeters squared
  Baseline: number analyzed (Participants) | 130
  Baseline | 1.0 (0.8)
  Discharge: number analyzed (Participants) | 120
  Discharge | 2.0 (0.6)
  3-6 Month: number analyzed (Participants) | 126
  3-6 Month | 1.8 (0.5)
  1 Year: number analyzed (Participants) | 117
  1 Year | 1.8 (0.6)
  2 Year: number analyzed (Participants) | 108
  2 Year | 1.6 (0.5)
  3 Year: number analyzed (Participants) | 100
  3 Year | 1.5 (0.5)
  4 Year: number analyzed (Participants) | 81
  4 Year | 1.5 (0.4)
  5 Year: number analyzed (Participants) | 89
  5 Year | 1.4 (0.5)

5. Secondary Outcome: Subject's New York Heart Association (NYHA) Functional Class Compared to Baseline.
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Symptoms of heart failure or the anginal syndrome may be present even at rest.
Time Frame: 3-6 Months and 1 through 5 Years compared to baseline
Population: This outcome is reported for subjects who received the Model 11000 surgical aortic heart valve where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
Participants
  Improve at 3-6 Months: number analyzed (Participants) | 128
  Improve at 3-6 Months | 89
  Same at 3-6 Months: number analyzed (Participants) | 128
  Same at 3-6 Months | 36
  Worse at 3-6 months: number analyzed (Participants) | 128
  Worse at 3-6 months | 3
  Improve at 1 Year: number analyzed (Participants) | 122
  Improve at 1 Year | 68
  Same at 1 Year: number analyzed (Participants) | 122
  Same at 1 Year | 48
  Worse at 1 Year: number analyzed (Participants) | 122
  Worse at 1 Year | 6
  Improve at 2 Years: number analyzed (Participants) | 111
  Improve at 2 Years | 68
  Same at 2 Years: number analyzed (Participants) | 111
  Same at 2 Years | 34
  Worse at 2 Years: number analyzed (Participants) | 111
  Worse at 2 Years | 9
  Improve at 3 Years: number analyzed (Participants) | 105
  Improve at 3 Years | 59
  Same at 3 Years: number analyzed (Participants) | 105
  Same at 3 Years | 41
  Worse at 3 Years: number analyzed (Participants) | 105
  Worse at 3 Years | 5
  Improve at 4 Years: number analyzed (Participants) | 101
  Improve at 4 Years | 55
  Same at 4 Years: number analyzed (Participants) | 101
  Same at 4 Years | 40
  Worse at 4 Years: number analyzed (Participants) | 101
  Worse at 4 Years | 6
  Improve at 5 Years: number analyzed (Participants) | 91
  Improve at 5 Years | 50
  Same at 5 Years: number analyzed (Participants) | 91
  Same at 5 Years | 33
  Worse at 5 Years: number analyzed (Participants) | 91
  Worse at 5 Years | 8

6. Secondary Outcome: Subject's Average Score at Baseline and 1 Year on the Quality of Life Survey
Description: The Medical Outcomes Study Short-Form 12 (SF-12) contains two components - the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
  The SF-12 Physical Component Summary questionnaire scale ranges from a maximum of 100, which reflects the best health status to a minimum of 0, which reflects the worst health status.
  The SF-12 Mental Component Summary scale ranges from a maximum of 100, which reflects the best health status to a minimum of 0, which reflects the worst health status.
Time Frame: Baseline and one year follow-up
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 56
units on a scale
  Physical Health - Baseline | 42.5 (10.2)
  Physical Health - 1 Year follow-up | 49 (7.4)
  Mental Health - Baseline | 50.2 (8.6)
  Mental Health - 1 Year follow-up | 51.2 (7.3)

7. Secondary Outcome: Subject's Average Score on the EQ-5D- Quality of Life Questionnaire Over Time
Description: The EQ-5D is a standardized questionnaire that asks subjects to rate themselves (no problems, some problems, extreme problems) on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale is indexed and ranges from a minimum of 0.275 and a maximum of 1.000. A lower number indicates the participants experiences more problems and a higher number indicates the participants experiences fewer problems.
Time Frame: Baseline and 1 Year
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 56
units on a scale
  Baseline | 0.81 (0.20)
  1 Year follow-up | 0.87 (0.20)

8. Other Pre Specified Outcome: Subject's Average White Blood Cell Count
Description: Laboratory analysis of White Blood Cell Count on blood drawn from subject; WBC fight infection.
Time Frame: Baseline, 3-6 Months, and 1 through 5 Years
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliters
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
10^3 cells/microliters
  Baseline | 7.0 (1.7)
  3-6 Months: number analyzed (Participants) | 124
  3-6 Months | 7.5 (2.2)
  1 Year: number analyzed (Participants) | 106
  1 Year | 7.3 (1.8)
  2 Year: number analyzed (Participants) | 108
  2 Year | 7.2 (1.6)
  3 Year: number analyzed (Participants) | 95
  3 Year | 7.1 (1.8)
  4 Year: number analyzed (Participants) | 80
  4 Year | 7.2 (1.8)
  5 Year: number analyzed (Participants) | 70
  5 Year | 7.2 (1.9)

9. Other Pre Specified Outcome: Subject's Average Red Blood Cells Count
Description: Laboratory Analysis of Red Blood Cell Count on blood drawn from subjects; RBC carry oxygen.
Time Frame: Baseline, 3-6 Months, and 1 through 5 Years
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliters
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
10^6 cells/microliters
  Baseline | 4.5 (0.5)
  3-6 Months: number analyzed (Participants) | 124
  3-6 Months | 4.7 (0.5)
  1 Year: number analyzed (Participants) | 106
  1 Year | 4.6 (0.4)
  2 Year: number analyzed (Participants) | 108
  2 Year | 4.6 (0.5)
  3 Year: number analyzed (Participants) | 95
  3 Year | 4.7 (0.5)
  4 Year: number analyzed (Participants) | 80
  4 Year | 4.6 (0.5)
  5 Year: number analyzed (Participants) | 70
  5 Year | 4.6 (0.5)

10. Other Pre Specified Outcome: Subject's Average Hemoglobin Count
Description: Laboratory Analysis of Hemoglobin Count on blood drawn from subjects. Hemoglobin is an oxygen-carrying protein in red blood cells.
Time Frame: Baseline, 3-6 months, and 1 through 5 years
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
g/dl
  Baseline | 13.5 (1.5)
  3-6 Months: number analyzed (Participants) | 124
  3-6 Months | 13.3 (1.4)
  1 Year: number analyzed (Participants) | 107
  1 Year | 13.7 (1.4)
  2 Years: number analyzed (Participants) | 108
  2 Years | 13.8 (1.5)
  3 Years: number analyzed (Participants) | 95
  3 Years | 14.0 (1.3)
  4 Years: number analyzed (Participants) | 80
  4 Years | 13.9 (1.6)
  5 Years: number analyzed (Participants) | 70
  5 Years | 13.7 (1.5)

11. Other Pre Specified Outcome: Subject's Average Hematocrit Percentage
Description: Laboratory Analysis of Hematocrit Percentage on blood drawn from subjects. Hematocrit is the proportion of red blood cells to the fluid component(plasma) in the blood.
Time Frame: Baseline, 3-6 Months, and 1 through 5 Years
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
percentage of red blood cells
  Baseline | 40.1 (4.2)
  3-6 Months: number analyzed (Participants) | 124
  3-6 Months | 40.5 (3.8)
  1 Year: number analyzed (Participants) | 106
  1 Year | 40.7 (3.5)
  2 Years: number analyzed (Participants) | 108
  2 Years | 41.1 (3.7)
  3 Years: number analyzed (Participants) | 95
  3 Years | 41.9 (3.6)
  4 Years: number analyzed (Participants) | 80
  4 Years | 41.9 (7.0)
  5 Years: number analyzed (Participants) | 70
  5 Years | 41.4 (4.0)

12. Other Pre Specified Outcome: Subject's Average Platelet Count
Description: Laboratory Analysis of Platelet Count on blood drawn from subjects; platelets help with blood clotting.
Time Frame: Baseline, 3-6 Months, and 1 through 5 Years
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: 10^3 platelets per microliter
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
10^3 platelets per microliter
  Baseline | 196.0 (48.3)
  3-6 Months: number analyzed (Participants) | 124
  3-6 Months | 203.1 (55.9)
  1 Year: number analyzed (Participants) | 106
  1 Year | 196.6 (49.8)
  2 Years: number analyzed (Participants) | 108
  2 Years | 195.8 (47.1)
  3 Years: number analyzed (Participants) | 95
  3 Years | 188.7 (45.4)
  4 Years: number analyzed (Participants) | 80
  4 Years | 194.4 (54.8)
  5 Years: number analyzed (Participants) | 70
  5 Years | 206.6 (57.7)

13. Other Pre Specified Outcome: Subject's Average Plasma Free Hemoglobin
Description: Laboratory Analysis of Plasma Free Hemoglobin on blood drawn from subjects. This blood test measures the level of free hemoglobin in the liquid part of the blood (the serum).
Time Frame: Baseline, 3-6 Months, and 1 through 5 Years
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
mg/dl
  Baseline: number analyzed (Participants) | 51
  Baseline | 12.9 (13.9)
  3-6 Years: number analyzed (Participants) | 101
  3-6 Years | 12.1 (8.1)
  1 Year: number analyzed (Participants) | 75
  1 Year | 14.2 (24.6)
  2 Years: number analyzed (Participants) | 108
  2 Years | 18.6 (27.7)
  3 Years: number analyzed (Participants) | 97
  3 Years | 19.3 (25.7)
  4 Years: number analyzed (Participants) | 75
  4 Years | 20.1 (26.6)
  5 Years: number analyzed (Participants) | 70
  5 Years | 28.1 (38.5)

14. Other Pre Specified Outcome: Subject's Average Serum Creatinine
Description: Laboratory Analysis of Serum Creatinine on blood drawn from subjects. Creatinine blood test is a test that measures kidney function.
Time Frame: Baseline
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: micromol/l
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 53
micromol/l | 84.0 (17.4)

15. Other Pre Specified Outcome: Subject's Average International Normalized Ratio
Description: Laboratory Analysis of International Normalized Ratio (INR) on blood drawn from subjects.
  The INR is a calculation based on results of a prothrombin time (PT). The PT is a blood test that measures the time it takes for the liquid portion (plasma) of the blood to clot.
Time Frame: Baseline, Discharge, 3-6 Months, 1 Year, 3 Years, and 5 Years
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
Ratio
  Baseline | 1.0 (0.1)
  Discharge: number analyzed (Participants) | 112
  Discharge | 1.9 (1.0)
  3-6 Months: number analyzed (Participants) | 123
  3-6 Months | 1.9 (0.8)
  1 Year: number analyzed (Participants) | 106
  1 Year | 1.2 (0.5)
  3 Years: number analyzed (Participants) | 96
  3 Years | 1.2 (0.6)
  5 Years: number analyzed (Participants) | 69
  5 Years | 1.2 (0.6)

16. Other Pre Specified Outcome: Subject's Average Partial Thromboplastin Time
Description: Laboratory Analysis of partial thromboplastin time (PTT) on blood drawn from subjects. PTT is a blood test that looks at how long it takes for the blood to clot.
Time Frame: Baseline, Discharge, 3-6 Months, 1 Year, 3 Years, and 5 Years
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
Seconds
  Baseline: number analyzed (Participants) | 132
  Baseline | 30.0 (6.5)
  Discharge: number analyzed (Participants) | 108
  Discharge | 39.5 (10.5)
  3-6 Months: number analyzed (Participants) | 121
  3-6 Months | 35.1 (8.9)
  1 Year: number analyzed (Participants) | 106
  1 Year | 28.6 (5.2)
  3 Years: number analyzed (Participants) | 94
  3 Years | 29.9 (10.2)
  5 Years: number analyzed (Participants) | 69
  5 Years | 33.6 (10.2)

17. Other Pre Specified Outcome: Subject's Average Prothrombin Time
Description: Laboratory Analysis of Prothrombin Time (PT) on blood drawn from subjects. The PT is a blood test that measures the time it takes for the liquid portion (plasma) of the blood to clot.
Time Frame: Baseline, Discharge, 3-6 Months, 1 Year, 3 Years, and 5 Years
Population: This outcome is reported for subjects who received a Model 11000 surgical aortic heart valve where data is available.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Aortic Bioprosthesis, Model 11000
Number analyzed (Participants) | 133
Seconds
  Baseline: number analyzed (Participants) | 113
  Baseline | 11.9 (1.9)
  Discharge: number analyzed (Participants) | 112
  Discharge | 21.5 (11.5)
  3-6 Months: number analyzed (Participants) | 104
  3-6 Months | 19.4 (9.1)
  1 Year: number analyzed (Participants) | 88
  1 Year | 14.0 (5.9)
  3 Years: number analyzed (Participants) | 79
  3 Years | 13.4 (5.3)
  5 Years: number analyzed (Participants) | 58
  5 Years | 12.5 (4.3)

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through five years post implant
Arm/Group | Aortic Bioprosthesis, Model 11000
All-Cause Mortality (participants affected / at risk) | 21/133
Serious Adverse Events (participants affected / at risk) | 74/133
Other Adverse Events (participants affected / at risk) | 41/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortic Bioprosthesis, Model 11000 (N=133)
Anemia - non-bleeding related (Blood and lymphatic system disorders) | 1 (1)
Angina, stable (Cardiac disorders) | 1 (1)
Arrhythmia-AV block III (Cardiac disorders) | 1 (1)
Arrhythmia - AV block - 3rd degree (Cardiac disorders) | 3 (3)
Arrhythmia - bradycardia (Cardiac disorders) | 1 (1)
Arrhythmia - paroxysmal atrial fibrillation (PAF) (Cardiac disorders) | 7 (9)
Arrhythmia - persistent atrial fibrillation (Cardiac disorders) | 3 (4)
Arrhythmia - supraventricular tachycardia (SVT) (Cardiac disorders) | 1 (1)
Arrhythmia - tachy-bradycardia (Cardiac disorders) | 1 (1)
Arrhythmia - ventricular fibrillation (Cardiac disorders) | 1 (1)
Biliary (gallbladder) (Gastrointestinal disorders) | 3 (4)
Bleeding event (Blood and lymphatic system disorders) | 12 (12)
Bone fracture/break (Musculoskeletal and connective tissue disorders) | 3 (3)
Cancer - newly diagnosed (General disorders) | 6 (6)
Cancer - progression of underlying disease (General disorders) | 2 (5)
Cardiac arrest (Cardiac disorders) | 3 (3)
Cardiac decompensation (Cardiac disorders) | 4 (4)
Cardiovascular - other (Cardiac disorders) | 2 (2)
Cardiovascular - other --> infection inflammation (Cardiac disorders) | 1 (1)
Endocarditis (Cardiac disorders) | 1 (1)
Endocrine complications (Endocrine disorders) | 1 (1)
Gastrointestinal - other (Gastrointestinal disorders) | 5 (6)
Genitourinary - other (Renal and urinary disorders) | 2 (3)
Heart failure - chronic (CHF) (Cardiac disorders) | 2 (2)
Hypertension - systemic (Cardiac disorders) | 1 (1)
Muscular skeletal / dermatologic - other (Musculoskeletal and connective tissue disorders) | 5 (6)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nonspecific, unknown or other body system - other complication (General disorders) | 4 (5)
Pancreatic complication (Gastrointestinal disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericardial effusion - major (Cardiac disorders) | 4 (4)
Pericardial effusion - minor (Cardiac disorders) | 1 (1)
Pericardial tamponade - major (Cardiac disorders) | 3 (3)
Pleural effusion - bilateral (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion - left (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion - right (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/respiratory - other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal - other (Renal and urinary disorders) | 3 (3)
Renal dysfunction (Renal and urinary disorders) | 1 (1)
Renal failure - acute (Renal and urinary disorders) | 2 (2)
Renal failure - chronic (Renal and urinary disorders) | 1 (1)
Respiratory dysfunction/insufficiency (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure - pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory infection - pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory infection - upper (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sternal wound/thoracic infection (Musculoskeletal and connective tissue disorders) | 4 (4)
Sudden death (General disorders) | 1 (1)
Tachy-bradycardia (Cardiac disorders) | 1 (1)
Thromboembolism (Cardiac disorders) | 5 (5)
Transient psychotic syndrome (Psychiatric disorders) | 1 (1)
Valve thrombosis (Cardiac disorders) | 1 (1)
Vascular - other (Vascular disorders) | 3 (3)
Vision disorder (Eye disorders) | 1 (1)
Wound infection - other (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortic Bioprosthesis, Model 11000 (N=133)
Arrhythmia - AV block - 1st degree (Cardiac disorders) | 1 (1)
Arrhythmia - paroxysmal atrial fibrillation (PAF) (Cardiac disorders) | 18 (18)
Arrhythmia - paroxysmal atrial tachycardia (PAT) (Cardiac disorders) | 1 (1)
Arrhythmia - permanent atrial fibrillation (Cardiac disorders) | 1 (1)
Arrhythmia - persistent atrial fibrillation (Cardiac disorders) | 4 (4)
Arrhythmia - tachy-bradycardia (Cardiac disorders) | 1 (1)
Bleeding event (Blood and lymphatic system disorders) | 1 (1)
Cardiovascular - other (Cardiac disorders) | 1 (1)
Non structural valve dysfunction (Cardiac disorders) | 1 (1)
Nonspecific, unknown or other body system - other complication (General disorders) | 1 (1)
Pericardial effusion - minor (Cardiac disorders) | 1 (1)
Pleural effusion - right (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Renal dysfunction (Renal and urinary disorders) | 2 (2)
Respiratory infection - upper (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stenosis - tricuspid - moderate (Cardiac disorders) | 1 (1)
Transient psychotic syndrome (Psychiatric disorders) | 3 (3)
Vision disorder (Eye disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can't publish/present on overall study results not yet published but may publish his own data subject to EW review prior to submission/presentation, but data analyses of site-specific results can occur only in intervals as specified in the CTA. Publication/presentation of the PI's site-specific results of devices which haven't been market released and which still may be undergoing development, shall not include claims of device safety/effectiveness and will require the review/approval of EW.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-05-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT01651052/Prot_SAP_000.pdf